CLINICAL TRIAL: NCT05446623
Title: Comparative Study of General Anesthesia With or Without Opioid on the Cardiac Index During Total Hip Arthroplasty
Brief Title: Cardiac Index and General Anesthesia Without Opioid.
Acronym: OFFLOW
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Montauban (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2020-A02873-36
Record Dates: First submitted 2022-06-19; First posted 2022-07-06 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hip Arthropathy; Hip Disease
Keywords: cardiac index; total hip arthroplasty; opioid free anesthesia
MeSH Terms: interventions — Dexmedetomidine; Sufentanil

STUDY DESIGN:
Intervention Model Description: It is a monocentric, randomized study comparing two strategies of general anesthesia for programmed total hip arthroplasty.
  Patients who gave their consent for the study during the anesthesia consultation, will be randomized into two groups depending on the type of general anesthesia: Opioid free anesthesia (OFA), or anesthesia with opioid (OA) The patients included in the OFA group will receive a bolus of Dexmedethomidine at the beginning of the surgery. The one in the OA group will be given a bolus of Sufentanil before and during the surgery. When the specific sequence will be completed, the care of all the patient will return to usual.
  During the anesthesia induction and during the surgery cardiovascular data will be collected. The cardiac index will be measured thanks to a non invasive cardiac monitoring called NICCOMO® (v3.5.2).
Who Masked: Participant, Investigator
Masking Description: Randomized into two groups depending on the type of general anesthesia: Opioid free anesthesia (OFA), or anesthesia with opioid (OA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid free anesthesia (OFA) (Active Comparator): The patients included in the OFA group will receive a bolus of Dexmedetomidine at the beginning of the surgery.
  Interventions: Drug: Dexmedetomidine
- anesthesia with opioid (OA) (Sham Comparator): The one in the OA group will be given a bolus of Sufentanil before and during the surgery. When the specific sequence will be completed, the care of all the patient will return to usual.
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Dexmedetomidine — Opioid free anesthesia (OFA) consists in the simultaneous administration of alpha2-agonist (for example the dexmedetomidine), sodium channel blocker (lidocaine), and NMDA antagonists receptors (Ketamine). Its aim is to control de cardiovascular nociceptive response to the surgical stimulation.
  Other Names: DEXDOR
  Arms: Opioid free anesthesia (OFA)
Drug: Sufentanil — The one in the OA group will be given a bolus of Sufentanil before and during the surgery.
  Other Names: Sufenta
  Arms: anesthesia with opioid (OA)

SUMMARY:
General anesthesia used to be based on the association of hypnotics and opioid drugs. But recent studies showed that opioids may be related to a many different complications, like respiratory distress, hyperalgesia.

Opioid free anesthesia (OFA) aim is to control de cardiovascular nociceptive response to the surgical stimulation. The scientific literature is not clear yet on the cardiovascular effect of the OFA. Optimization of the cardiac index proved its worth in reducing morbidity and mortality.

The purpose of this study is to increase our understanding of the impact of opioid free anesthesia on the cardiovascular system and to evaluate the effectiveness and the security of the technic.

DETAILED DESCRIPTION:
General anesthesia used to be based on the association of hypnotics and opioid drugs. But recent studies showed that opioïds may be related to a many different complications, like respiratory distress, hyperalgesia etc… Those sides effects are known, but there might be some recent technics that could allow anesthesiologist to reduce those unintended symptoms. As surgery became an important pilar of the modern medicine even in fragile people, the weight of opioids sides effect increased.

Opioid free anesthesia (OFA) consists in the simultaneous administration of alpha2-agonist (for example the dexmedetomidine (DEXDOR)), sodium channel blocker (lidocaine), and N-methyl-D-aspartate (NMDA) antagonists receptors (Ketamine). Its aim is to control de cardiovascular nociceptive response to the surgical stimulation. The scientific literature is not clear yet on the cardiovascular effect of the OFA. Optimization of the cardiac index proved its worth in reducing morbidity and mortality. The investigators thinks that exploring the impact of two different general anesthesia technics on cardiac index, might allow anesthesiologists to have a better understanding of the anesthetic strategy applied to the patient.

General anesthesia with or without opioid is used on a daily basis at the hospital center of Montauban. The possible sides effects of OFA as well as those affiliate to balanced anesthesia are known by all the care workers.

The purpose of this study is to increase our understanding of the impact of opioid free anesthesia on the cardiovascular system and to evaluate the effectiveness and the security of the technic.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients for scheduled total hip arthroplasty with general anesthesia.
* Patients with an American Society of Anesthesiologists (ASA) score between 1 and 3
* Patient who has received appropriate information and has provided informed consent.
* Patient with French social security system.

Exclusion Criteria:

* Patients eligible to rapid sequence intubation.
* Patients with medical contraindication to the use of OFA : allergy to one of the drug used in the protocol, spontaneous bradycardia under 40bpm or atrioventricular block.
* Patients with a medical condition that could alter measurement of cardiac index by NICCOMO™: acute pulmonary oedema, severe valvular heart disease, pulmonary hypertension, atrial fibrillation.
* Patients who cannot give their informed consent.
* Patients pregnant or breastfeeding.
* Patients odler than 90 years old or with a weigh superior at 150kg.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-10-02 (Estimated); Study Completion 2024-01-02 (Estimated)

PRIMARY OUTCOMES:
the impact of opioid free anesthesia on the cardiac index | 60 minutes
  The main objective of this study is to evaluate the impact of opioid free anesthesia on the cardiac index and comparing it to the general anesthesia protocol with opioids.

SECONDARY OUTCOMES:
Assess the impact of the OFA in hemodynamical state | 60 minutes
  To assess the impact of the OFA protocol on Blood pressure (variation of Blood pressure measured in mmHg)
Assess the impact of the OFA protocol on heart rate | 60 minutes
  To assess the impact of the OFA protocol on heart rate (variation in heart rate measured in beats per minute)
Assess the impact of OFA on postoperative pain | 48 hours
  To assess the impact of OFA on postoperative pain (variation in numeric rating scales) From 0 to 10 => Zero represents "no pain," whereas 10 represents the opposite end of the pain continuum (e.g., "the most intense pain imaginable," "pain as intense as it could be," "maximum pain").
Assess the impact of OFA on the consumption of postoperative morphine | 48 hours
  To assess the impact of OFA on the consumption of postoperative morphine (consumption in mg)

CONTACTS AND LOCATIONS:
Locations (1):
- Edmundo Pereira de Souza Neto, Montauban, Tarn Et Garonne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Background] Yi P, Pryzbylkowski P. Opioid Induced Hyperalgesia. Pain Med. 2015 Oct;16 Suppl 1:S32-6. doi: 10.1111/pme.12914. PMID 26461074
- [Background] Lavand'homme P, Estebe JP. Opioid-free anesthesia: a different regard to anesthesia practice. Curr Opin Anaesthesiol. 2018 Oct;31(5):556-561. doi: 10.1097/ACO.0000000000000632. PMID 29994942
- [Background] Mauermann E, Ruppen W, Bandschapp O. Different protocols used today to achieve total opioid-free general anesthesia without locoregional blocks. Best Pract Res Clin Anaesthesiol. 2017 Dec;31(4):533-545. doi: 10.1016/j.bpa.2017.11.003. Epub 2017 Nov 24. PMID 29739542
- [Background] Mulier JP. Is opioid-free general anesthesia for breast and gynecological surgery a viable option? Curr Opin Anaesthesiol. 2019 Jun;32(3):257-262. doi: 10.1097/ACO.0000000000000716. PMID 31045633
- [Background] Beloeil H. Opioid-free anesthesia. Best Pract Res Clin Anaesthesiol. 2019 Sep;33(3):353-360. doi: 10.1016/j.bpa.2019.09.002. Epub 2019 Sep 26. PMID 31785720
- [Background] Chia PA, Cannesson M, Bui CCM. Opioid free anesthesia: feasible? Curr Opin Anaesthesiol. 2020 Aug;33(4):512-517. doi: 10.1097/ACO.0000000000000878. PMID 32530891
- [Background] Bugada D, Lorini LF, Lavand'homme P. Opioid free anesthesia: evidence for short and long-term outcome. Minerva Anestesiol. 2021 Feb;87(2):230-237. doi: 10.23736/S0375-9393.20.14515-2. Epub 2020 Aug 4. PMID 32755088
- [Background] Lavand'homme P, Steyaert A. Opioid-free anesthesia opioid side effects: Tolerance and hyperalgesia. Best Pract Res Clin Anaesthesiol. 2017 Dec;31(4):487-498. doi: 10.1016/j.bpa.2017.05.003. Epub 2017 May 17. PMID 29739537
- [Background] Kharasch ED, Clark JD. Opioid-free Anesthesia: Time to Regain Our Balance. Anesthesiology. 2021 Apr 1;134(4):509-514. doi: 10.1097/ALN.0000000000003705. No abstract available. PMID 33630018
- [Background] Forget P. Opioid-free anaesthesia. Why and how? A contextual analysis. Anaesth Crit Care Pain Med. 2019 Apr;38(2):169-172. doi: 10.1016/j.accpm.2018.05.002. Epub 2018 Sep 13. PMID 29775728
- [Background] Bakan M, Umutoglu T, Topuz U, Uysal H, Bayram M, Kadioglu H, Salihoglu Z. Opioid-free total intravenous anesthesia with propofol, dexmedetomidine and lidocaine infusions for laparoscopic cholecystectomy: a prospective, randomized, double-blinded study. Braz J Anesthesiol. 2015 May-Jun;65(3):191-9. doi: 10.1016/j.bjane.2014.05.001. Epub 2014 Jun 3. PMID 25925031
- [Background] Tempe DK, Sawhney C. Opioid-Free Anesthesia for Thoracic Surgery: A Step Forward. J Cardiothorac Vasc Anesth. 2020 Nov;34(11):3041-3043. doi: 10.1053/j.jvca.2020.07.022. Epub 2020 Jul 10. No abstract available. PMID 32739086
- [Background] Siu EY, Moon TS. Opioid-free and opioid-sparing anesthesia. Int Anesthesiol Clin. 2020 Spring;58(2):34-41. doi: 10.1097/AIA.0000000000000270. No abstract available. PMID 32004171
- [Background] Chakravarthy M. Opioid free cardiac anesthesia - A flash in the pan? Ann Card Anaesth. 2020 Apr-Jun;23(2):113-115. doi: 10.4103/aca.ACA_68_19. No abstract available. PMID 32275021
- See also: The Benefits of Opioid Free Anesthesia and the Precautions Necessary When Employing It. Transl Perioper Pain Med — http://www.transpopmed.org/articles/tppm/tppm-2019-7-104.php